CLINICAL TRIAL: NCT03748082
Title: Effects of Nitric Oxide on Vascular Responsiveness and on Endothelial Cells During Hemolysis in Patients With Pre-operative Endothelial Dysfunction Undergoing Prolonged Cardiopulmonary Bypass.
Brief Title: Effects of Nitric Oxide on the Endothelium During Hemolysis.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Spina, Stefano, M.D., Massachusetts General Hospital (Unknown); Marrazzo, Francesco, M.D., Massachusetts General Hospital (Unknown); Zadek, Francesco, M.D., Massachusetts General Hospital (Unknown); Jennifer En-Sian Ho M.D., Massachusetts General Hospital (Unknown); Naomi M Hamburg, M.D., Boston University (Unknown)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EndoNO
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Endothelial Dysfunction; Hemolysis Intravascular; Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Cardiac Surgery; Cardiopulmonary Bypass; Reactive Hyperemia Index; Nitric Oxide
MeSH Terms: conditions — Hemolysis; Cardiovascular Diseases | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Inhaled nitrogen will be administered via the cardiopulmonary bypass (CPB) machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the Intensive Care Unit (ICU). Test gas administration will commence at the onset of CPB and last for 24 hours.
  Interventions: Diagnostic Test: Reactive Hyperemia Index; Procedure: Endothelial Cells Collection
- Nitric Oxide (Experimental): Inhaled nitric oxide (iNO) will be administered via the CPB machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the ICU. Test gas administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, iNO will be weaned and discontinued.
  Interventions: Drug: Nitric Oxide; Diagnostic Test: Reactive Hyperemia Index; Procedure: Endothelial Cells Collection

INTERVENTIONS:
Drug: Nitric Oxide — Inhaled nitric oxide (iNO) will be administered via the CPB machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the ICU. Test gas administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, iNO will be weaned and discontinued.
  Other Names: iNO
  Arms: Nitric Oxide
Diagnostic Test: Reactive Hyperemia Index — Vascular responsiveness will be assessed with peripheral arterial tonometry which measures the transient increase in forearm blood flow (Reactive Hyperemia Index, RHI) in response to a five-minute occlusion of the brachial artery with a pressure cuff.
Procedure: Endothelial Cells Collection — Endothelial cells are collected before and after surgery from a peripheral vessel using a soft J-shaped wire inserted through an intravascular catheter.

SUMMARY:
This study is an ancillary (add-on) study to the clinical trial entitled "Effect of Nitric Oxide in Cardiac Surgery Patients With Endothelial Dysfunction", which has Clinical Trials.gov identifier NCT02836899. NCT02836899 trial randomizes cardiac surgical patients to receive either Nitric Oxide (NO) or a placebo during and after cardiac surgery.

This ancillary study aims to assess the effects of Nitric Oxide on vascular responsiveness and on endothelial function during hemolysis in patients with pre-operative endothelial dysfunction undergoing cardiac surgery requiring prolonged cardiopulmonary bypass.

DETAILED DESCRIPTION:
Endothelial cells regulate tissue perfusion by releasing nitric oxide (NO), a potent endogenous dilator of vascular smooth muscle cells, which modifies vascular tone. Under normal physiological conditions, vascular NO is released by endothelial NO synthase (eNOS). Impairment of the eNOS, as seen in patients with atherosclerosis, peripheral vascular disease, hypertension, obesity, and diabetes, is a feature of endothelial dysfunction.The inability to increment eNOS activity is particularly evident in conditions of decreased vascular NO bioavailability, such as during hemolysis associated with prolonged cardiopulmonary bypass (CPB>90 min). During hemolysis, ferrous plasma free hemoglobin (Oxy-Hb) is released into the circulation and can be injurious for the endothelial cells by exerting an oxidative and proinflammatory effect. Moreover, plasma free Oxy-Hb can scavenge vascular NO, reducing its bioavailability as ferrous Oxy-Hb is transformed into ferric methemoglobin (Met-Hb). The clinical results of reduced bioavailability of vascular NO have been found to be associated with both systemic and pulmonary vasoconstriction, ultimately leading to reduced tissue perfusion.

The exogenous administration of NO has been shown to prevent the scavenging of endogenous NO by inactivating the highly oxidative-reactive ferrous plasma Oxy-Hb to ferric Met-Hb. Our group is conducting a randomized controlled trial at Massachusetts General Hospital (Boston, USA) in patients with signs and symptoms of endothelial dysfunction, undergoing cardiac surgery requiring prolonged CPB and randomized to receive NO or placebo. However, the mechanisms underlying the beneficial systemic effects of NO administration have still to be determined. This is an ancillary study that aims to (I) assess the effects of hemolysis on vascular responsiveness and on endothelial function in patients with pre-operative endothelial dysfunction and (II) to determine the vascular protective effects of NO administration.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and randomized in the trial NCT02836899
* Provide written informed consent
* Age ≥ 18 years of age
* Elective cardiac or aortic surgery with CPB >90 minutes
* Clinical evidence of endothelial dysfunction assessed by a specifically designed questionnaire

Exclusion Criteria:

* Estimated Glomerular Filtration Rate less than 30 ml/min/1.73 m2
* Emergent cardiac surgery
* Life expectancy < 1 year at the time of enrollment
* Hemodynamic instability as defined by a systolic blood pressure <90 mmHg.
* Mean pulmonary artery pressure ≥ 40 mm Hg and PVR > 4 Wood Units.
* Left ventricular ejection fraction < 30% by echocardiography obtained within three months of enrollment
* Administration of one or more Packed Red Blood Cell (PRBC) transfusions in the week prior to enrollment
* X-ray contrast infusion less than 48 hours before surgery
* Evidence of hemolysis from any other origin:

  a. Intravascular: i. Intrinsic RBC defects leading to hemolytic anemia (eg, enzyme deficiencies, hemoglobinopathies, membrane defects) ii. Extrinsic: liver disease, hypersplenism, infections (eg, bartonella, babesia, malaria), treatment with oxidizing exogenous agents (eg, dapsone, nitrites, aniline dyes), exposure to other hemolytic agents (eg, lead, snake and spider bites), lymphocyte leukemia, autoimmune hemolytic disorders b. Extravascular: Infection (eg, clostridial sepsis, severe malaria), paroxysmal cold hemoglobinuria, cold agglutinin disease, paroxysmal nocturnal hemoglobinuria, iv infusion of Rho(D) immune globulin, iv infusion of hypotonic solutions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) | The test will be performed perioperatively before anesthesia induction and at 24 hours after CPB during ICU admission.
  A finger plethysmograph will measure the transient increase in forearm blood flow (Reactive Hyperemia Index, RHI) in response to a 5 minutes occlusion of the brachial artery with a pressure cuff (Peripheral Artery Tonometry).

OTHER OUTCOMES:
Endothelial Nitric Oxide Synthase (eNOS) enzymatic activity | Endothelial Cells will be collected perioperatively before anesthesia induction and at 24 hours after CPB during ICU admission.
  eNOS enzymatic activity will be measured in endothelial cells. Activation of eNOS will be assessed through quantification of its expression by quantitative immunofluorescence and through evaluation of phosphorylation levels at different enzymatic sites at baseline and in response to specific agonists; NO bioavailability will be evaluated through fluorescence intensity after challenge with agonists as A23187; additionally, nitrotyrosine levels and other markers will be measured to evaluate endothelial oxidative stress.
Pulmonary vascular resistances (PVR) | PVR will be measured every 6 hours after surgery for 24 hours after cardiopulmonary bypass start.
  PVR will be measured through a pulmonary artery catheter (PAC) placed in the internal jugular vein after induction of anesthesia. Cardiac output will be measured with the thermodilution technique and pulmonary vascular resistances will be calculated.
Systemic vascular resistances (SVR) | SVR will be measured every 6 hours after surgery for 24 hours after cardiopulmonary bypass start.
  SVR will be measured through a pulmonary artery catheter (PAC) placed in the internal jugular vein after induction of anesthesia. Cardiac output will be measured with the thermodilution technique and systemic vascular resistances will be calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lei C, Berra L, Rezoagli E, Yu B, Dong H, Yu S, Hou L, Chen M, Chen W, Wang H, Zheng Q, Shen J, Jin Z, Chen T, Zhao R, Christie E, Sabbisetti VS, Nordio F, Bonventre JV, Xiong L, Zapol WM. Nitric Oxide Decreases Acute Kidney Injury and Stage 3 Chronic Kidney Disease after Cardiac Surgery. Am J Respir Crit Care Med. 2018 Nov 15;198(10):1279-1287. doi: 10.1164/rccm.201710-2150OC. PMID 29932345
- [Background] Rezoagli E, Ichinose F, Strelow S, Roy N, Shelton K, Matsumine R, Chen L, Bittner EA, Bloch DB, Zapol WM, Berra L. Pulmonary and Systemic Vascular Resistances After Cardiopulmonary Bypass: Role of Hemolysis. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):505-515. doi: 10.1053/j.jvca.2016.06.009. Epub 2016 Jun 8. PMID 27590461
- [Background] Tabit CE, Shenouda SM, Holbrook M, Fetterman JL, Kiani S, Frame AA, Kluge MA, Held A, Dohadwala MM, Gokce N, Farb MG, Rosenzweig J, Ruderman N, Vita JA, Hamburg NM. Protein kinase C-beta contributes to impaired endothelial insulin signaling in humans with diabetes mellitus. Circulation. 2013 Jan 1;127(1):86-95. doi: 10.1161/CIRCULATIONAHA.112.127514. Epub 2012 Nov 30. PMID 23204109
- [Background] Hamburg NM, Keyes MJ, Larson MG, Vasan RS, Schnabel R, Pryde MM, Mitchell GF, Sheffy J, Vita JA, Benjamin EJ. Cross-sectional relations of digital vascular function to cardiovascular risk factors in the Framingham Heart Study. Circulation. 2008 May 13;117(19):2467-74. doi: 10.1161/CIRCULATIONAHA.107.748574. Epub 2008 May 5. PMID 18458169